CLINICAL TRIAL: NCT00284466
Title: Comparing Angiography: Multislice CT vs. Invasive Heart Catheterization (CACTI)
Brief Title: Comparing Angiography: Multislice CT Versus Invasive Heart Catheterization (CACTI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-IRB 2005-0377
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Arteriosclerosis
Keywords: coronary artery disease; cardiac catheterization; CT coronary angiography; coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MS-CT Coronary Angiography — MS-CT Coronary Angiography done

SUMMARY:
The purpose of the study is to compare the pictures of heart arteries obtained by MSCT scanner to the pictures obtained during heart catheterization. Our specific question is whether the MSCT scanner is accurate enough to replace heart catheterization in some situations for the evaluation of coronary heart disease.

DETAILED DESCRIPTION:
QUESTION: Compare the accuracy of multi-slice CT angiography (CTA) with invasive catheterization (Cath) in detecting and grading coronary lesions.

EXPERIMENTAL DESIGN: A prospective cohort analysis comparing the quantification of coronary atherosclerosis by Computed Tomographic angiography to that of invasive Catheterization. Subjects will be patients who are scheduled for non-urgent cardiac cath based on a clinical need to evaluate the coronary anatomy. Cath may be scheduled after a positive stress test or on the basis of concerning symptoms. If a patient consents to participation they will be scheduled for CTA no less than 3 and no more than 30 days prior to Cath. Comparison of lesions detected by the two imaging modalities in the proximal, mid and distal coronary arteries will be made. Grades of disease used will be the following 1). less than 50% 2). 50-75% 3). greater than 75% 4) Uninterpretable. Sensitivity and specificity will be calculated for CTA; in addition PPV and NPV will also be calculated. The 2 readers of the CTA will be blinded to the invasive angiography results. The 2 readers of the invasive angiography, who are blinded to the CTA results will be the standard of comparison. Analysis of data will be performed on a segmental, vessel, and patient basis.

POTENTIAL RISK: Risks associated with contrast exposure include the risk of allergic reaction and renal injury. There is a small risk of excessive bradycardia and hypotension with administration of metoprolol and nitroglycerine. CTA is associated with radiation exposure similar to the lower range of diagnostic catheterization.

POTENTIAL BENEFITS: No direct benefits are expected for the subjects of this study as the information will not be used to alter clinical decisions. Benefits to future patients may include the development of an non-invasive alternative to cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >18 years old with stable clinical symptoms who are scheduled for outpatient cardiac catheterization.
2. Able to provide written informed consent in accordance with the IRB.

Exclusion Criteria:

1. Symptoms of unstable angina/acute coronary syndrome
2. Known allergy or adverse reaction to CT radiocontrast and/or iodine.
3. Known absolute contraindication to Metoprolol.
4. Significant kidney disease including creatinine > 1.5 mg/dL or GFR < 60 ml/min.
5. Inability to breath-hold for up to 30 seconds.
6. Women who are Pregnant or Nursing
7. Atrial Fibrillation or any other arrhythmia that makes attaining a regular slow rhythm unlikely.
8. History of previous stent placement or coronary bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the ability of CTA to detect coronary disease of greater than 50% diameter stenosis (sensitivity, specificity, positive and negative predictive value) analyzed on a subject basis. | assess at time of CTA

SECONDARY OUTCOMES:
Assess CTA performance on both a vessel and coronary segment basis | assessed at time of CTA
Estimate the impact of coronary calcium score on ability to assess for coronary disease | assessed at time of CTA
Evaluate impact of scan quality of CTA performance measures | assessed at time of CTA

CONTACTS AND LOCATIONS:
Overall Officials: Jon G Keevil, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States